CLINICAL TRIAL: NCT05510921
Title: Evaluation of the Minimalist Music and Birdsongs in the Anxiety of Nursing Professionals in Oncology: a Randomized Clinical Trial
Brief Title: Evaluation of the Minimalist Music and Birdsongs in the Anxiety of Nursing Professionals in Oncology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Eliseth Ribeiro Leao, Senior research scientist, Hospital Israelita Albert Einstein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5483730
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Anxiety Disorders and Symptoms
Keywords: Nursing professionals; Anxiety; Oncology; Music; Nature
MeSH Terms: conditions — Anxiety Disorders; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): The control group will not receive any intervention
- Minimalist music group (Experimental): a live session of minimalist music piano piece
  Interventions: Other: Minimalist music group
- Minimalist music plus birdsongs group (Experimental): a live session of minimalist music piano piece with the superposition of bird song sounds
  Interventions: Other: Minimalist music + birdsongs group

INTERVENTIONS:
Other: Minimalist music group — Participants in this group will listen individually a live session of minimalist music piano piece, in a break room in the oncology sector, lasting between 10 and 15 minutes.
  Arms: Minimalist music group
Other: Minimalist music + birdsongs group — Participants in this group will listen individually a live session of minimalist music piano piece with the superposition of bird song sounds, in a break room in the oncology sector, lasting between 10 and 15 minutes.
  Arms: Minimalist music plus birdsongs group

SUMMARY:
This project aims to investigate the effects of an intervention involving minimalist piano music and bird singing on the anxiety of nursing professionals working in the Oncology sector of a hospital.

DETAILED DESCRIPTION:
The demand for care with mental health of nursing professionals is increasingly present, considering the high rate of anxiety symptoms presented by the teams providing health care within hospitals. Oncology is one of the sectors where professionals have constant contact with situations of suffering and death, being a place where the enlargement of therapeutic tools for handling anxiety symptoms may bring benefits. Scientific literature has never described the effectiveness of works with minimalist music and birds singing used simultaneously with anxiety relief resources. Objective: Assess the effects of music intervention, with minimalist repertoire, with or without association to birds singing over anxiety of nursing professionals that work in Oncology. Method: Randomized Clinical controlled trial. The study will be performed in the Oncology sector of Israeli Hospital Albert Einstein located in São Paulo, Brazil and the population consists in 100 nursing professionals. The intervention will consist in a musical part, especially developed for this study and in recording of birds singing, played live for each one of the participants, individually with 10 to 15 minutes duration. The instrument for anxiety assessment chosen for this project is short-form of state-trait anxiety inventory (STAI-S-6). The project was approved by the research ethics committee, whose identification number on Plataforma Brasil (CAAE) is 59498222.6.0000.0071

ELIGIBILITY:
Inclusion Criteria:

* Nursing professionals working in oncology Unit
* Over 18 years old

Exclusion Criteria:

* Nursing professionals who, for whatever reason, are unable to fully participate of the proposed musical intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline levels of anxiety at immediately post intervention | immediately pre intervention and immediately post intervention.
  To assess the anxiety of the study participant, the reduced scale of trait anxiety (STAI-S-6), validated in Brazil in a large sample of Brazilians, will be used. There are 6 questions that assess how the individual is feeling at the present moment and can be answered with 4 options on a 4-point Likert scale: 1- almost never; 2- sometimes; 3- frequently; 4- almost always. This gives a score range from 6 to 24. To create scores compatible with the original STAI-S scores, the STAI-6 scores will be divided by 6 and multiplied by 20 to give a range from 20 to 80.STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).

CONTACTS AND LOCATIONS:
Overall Officials: Eliseth R Leão, PhD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leao ER, Dal Fabbro DR, Oliveira RB, Santos IR, Victor ED, Aquarone RL, Andrade CB, Ribeiro VF, Oliveira RC, Friedlander R, Ferreira DS. Stress, self-esteem and well-being among female health professionals: A randomized clinical trial on the impact of a self-care intervention mediated by the senses. PLoS One. 2017 Feb 27;12(2):e0172455. doi: 10.1371/journal.pone.0172455. eCollection 2017. PMID 28241070

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/21/NCT05510921/Prot_ICF_000.pdf